CLINICAL TRIAL: NCT04669119
Title: Effects of Bromelain and Boswellia Serrata Casperome With Centella Asiatica and Thiamine, Riboflavin, Pyridoxine, Vitamin D, Superoxide Dismutase on Edema, Paresthesia and Postoperative Pain After Quadrantectomy With or Without Sentinel Lymph Node Biopsy: Blinded Randomized Controlled Study
Brief Title: Effects of Bromelain and Boswellia Serrata Casperome With Centella Asiatica and Vitamins on Edema, Paresthesia and Postoperative Pain After Quadrantectomy With or Without Sentinel Lymph Node Biopsy.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Angela Gurrado, Prof., University of Bari Aldo Moro
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020/6422
Record Dates: First submitted 2020-12-01; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer Female; Pain, Postoperative
Keywords: Dietary Supplements; Breast Cancer; Postoperative pain; Postoperative edema; Postoperative collections
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms | interventions — Bromelains; Centella asiatica extract; Vitamins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bromelain/Boswellia Serrata Casperome and Centella Asiatica/Vitamins (Experimental): Patients treated post-operatively for 30 days with Bromelain/Boswellia Serrata Casperome and Centella Asiatica/Vitamins
  Interventions: Dietary Supplement: Bromelain/Boswellia Serrata Casperome; Dietary Supplement: Centella Asiatica/Vitamins
- Bromelain/Boswellia Serrata Casperome and placebo (Experimental): Patients treated post-operatively for 30 days with Bromelain/Boswellia Serrata Casperome and placebo
  Interventions: Dietary Supplement: Bromelain/Boswellia Serrata Casperome; Dietary Supplement: Placebo
- Placebo (Placebo Comparator): Patients treated post-operatively for 30 days with placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bromelain/Boswellia Serrata Casperome — Dietary supplement already commercialized based on Bromelain/Boswellia Serrata Casperome (Arm A and B), called Siben by Agaton
  Arms: Bromelain/Boswellia Serrata Casperome and Centella Asiatica/Vitamins; Bromelain/Boswellia Serrata Casperome and placebo
Dietary Supplement: Centella Asiatica/Vitamins — Dietary supplement already commercialized based on Centella Asiatica/Vitamins (Arm B), called Kardinal V by Agaton
  Arms: Bromelain/Boswellia Serrata Casperome and Centella Asiatica/Vitamins
Dietary Supplement: Placebo — Placebo
  Arms: Bromelain/Boswellia Serrata Casperome and placebo; Placebo

SUMMARY:
Aim: to investigate the effects of dietary supplements on postoperative edema and pain in patients undergoing quadrantectomy for breast cancer.

Methods: 120 patients will be randomized into 3 groups: A, treated with Bromelain/Boswellia Serrata Casperome and Centella Asiatica with Vitamins for 30 days; B, treated with Bromelain/Bosswellia Serrata and placebo for 30 days; C, treated with 2 placebos. Inclusion criteria: adult (>18 years) patients with breast cancer undergoing quadrantectomy with or without sentinel lymph node biopsy. Exclusion criteria: diabetic neuropathy, previous breast/chest surgeries, allergies to studied drugs, severe kidney failure, alcohol and toxics addiction, axillary lymphadenectomy. Patients will be studied through ultrasound examination for edema and collections, VAS and DN4 for pain, during 30 postoperative days. Patients will also be studied through psychological and physiatric evaluations. Wilcoxon, T student, Chi-Squared tests will be used to evaluate the outcomes. STATA 14 (StataCorp LP, College Station, Tex, USA) will be used for the analysis. P<0.05 will be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years) with breast cancer undergoing quadrantectomy with or without sentinel lymph node biopsy

Exclusion Criteria:

* Diabetical neuropathy
* Previous breast/chest surgery
* Allergies to studied drugs
* Severe kidney failure
* Alcohol and toxics addiction
* Axillary lymphadenectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-12-31 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in postoperative normalized echogenicity of breast and subcutaneous tissue from the first to the 30th day after quadrantectomy with or without sentinel lymph node biopsy | 30 days
  Ultrasound measured postoperative edema, obtained through the evaluation of normalized echogenicity, of breast and subcutaneous tissue after quadrantectomy with or without sentinel lymph node biopsy

SECONDARY OUTCOMES:
Number of participants with postoperative fluid collections in the breast and or subcutaneous tissue during 30 days after quadrantectomy with or without sentinel lymph node biopsy | 30 days
  Ultrasound measured postoperative collections of breast and subcutaneous tissue after quadrantectomy with or without sentinel lymph node biopsy
Change in postoperative pain measured daily through VAS (visual analogue scale) from the first to the 30th day after quadrantectomy with or without sentinel lymph node biopsy | 30 days
  VAS (visual analogue scale) from 0 (absence of pain) to 10 (worst pain)
Change in postoperative probability of neuropathic pain measured daily through DN4 (Douleur Neuropathique en 4 Questions) from the first to the 30th day after quadrantectomy with or without sentinel lymph node biopsy | 30 days
  DN4 (Douleur Neuropathique en 4 Questions) from 0 (low probability of neuropathic pain) to 10 (high probability of neuropathic pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: No